CLINICAL TRIAL: NCT02610972
Title: Assessing the Usability and Clinical Utility of the Congo Red Dot Test: A Case-control Study
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: 4005A
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Preeclampsia
Keywords: Congo Red test GV-005
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CLINICALLY CONFIRMED PREECLAMPSIA: Women clinically diagnosed with preeclampsia (severe, mild or superimposed) during pregnancy will provide a urine sample in the postpartum period to determine the presence or absence of proteinuria using the Congo Red test GV-005.
  Interventions: Device: Congo Red test GV-005
- CLINICALLY HEALTHY: Women with a delivery of a healthy normal baby at term (induction of labor or an elective Caesarean Section) will provide a urine sample in the postpartum period to determine the presence or absence of proteinuria using the Congo Red test GV-005.
  Interventions: Device: Congo Red test GV-005

INTERVENTIONS:
Device: Congo Red test GV-005 — Congo Red test GV-005 test is a simple test has been developed to detect unfolded or misfolded proteins in urine.

SUMMARY:
A case-control study will evaluate the clinical utility of the Congo Red test GV-005 in following women with a clinical diagnosis of preeclampsia and clinically healthy women in the postpartum period

DETAILED DESCRIPTION:
A case-control study (n=150) will evaluate the clinical utility of the Congo Red test GV-005 in following women with a clinical diagnosis of preeclampsia and clinically healthy women in the postpartum period. Women with preeclampsia (n=100) (cases) and clinically healthy women (n=50)(controls) who are hospitalized postpartum will be recruited for the trial. All women will be asked to provide a urine sample. Samples will be collected daily during a woman's hospitalization. The Congo Red test GV-005 and a standard urine dipstick proteinuria test will be performed by a lab technician within 72 hours of sample collection. The purpose of this research is to evaluate progression of urine congophilia postpartum by following patients diagnosed with preeclampsia and clinically healthy women.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum
* Clinical diagnosis of preeclampsia (severe, mild or superimposed) including eclampsia (n=100) OR Clinically healthy (n=50)
* Eligible to consent for research
* Agree to comply with study procedures
* Able to give informed consent

Exclusion Criteria:

* None

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women attending Dhaka Medical College (Dhaka) with clinically confirmed cases of preeclampsia and clinically healthy women who deliver at term will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, Dr, Principal Investigator — Gynuity Health Projects
Locations (2):
- Dhaka Medical College, Dhaka, Bangladesh
- Hospital Materno-Infantil Inguarán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CLINICALLY CONFIRMED PREECLAMPSIA | CLINICALLY HEALTHY
Started | 100 | 50
Completed | 100 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLINICALLY CONFIRMED PREECLAMPSIA | CLINICALLY HEALTHY | Total
Number analyzed (Participants) | 100 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.86 (5.34) | 24.82 (5.08) | 24.85 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 50 | 150
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Bangladesh | 100 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Urine Congophilia Using Congo Red Test GV-005
Description: Prevalence of urine congophilia using Congo Red test GV-005
Time Frame: within 72 hours of urine sample collection
Measure: Count of Participants; unit: Participants
Arm/Group | CLINICALLY CONFIRMED PREECLAMPSIA | CLINICALLY HEALTHY
Number analyzed (Participants) | 100 | 50
Participants | 87 | 18

ADVERSE EVENTS:
Time Frame: 72 hours from time of enrollment
Arm/Group | CLINICALLY CONFIRMED PREECLAMPSIA | CLINICALLY HEALTHY
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/50
Other Adverse Events (participants affected / at risk) | 0/100 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT02610972/Prot_SAP_000.pdf